CLINICAL TRIAL: NCT05610059
Title: Improving Hypertension Medication Adherence for Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: R01NR018469 (NIH)
Record Dates: First submitted 2022-10-25; First posted 2022-11-09 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Aging; Medication Adherence; Hypertension
MeSH Terms: conditions — Medication Adherence; Hypertension

STUDY DESIGN:
Intervention Model Description: Participants will be screened and assigned to one of two groups using a blood pressure technology system.
Who Masked: Participant, Outcomes Assessor
Masking Description: All primary and secondary outcomes completed at 3-months and 6-months are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood Pressure Technology System M (Other): These participants will receive information about high blood pressure, medications and strategies that can be used to take medications and manage blood pressure. They will complete a mid-assessment at 3-months and a post-assessment at 6-months.
  Interventions: Other: Blood Pressure Technology System M
- Blood Pressure Technology System E (Other): These participants receive information about high blood pressure and medications. They will complete a mid-assessment at 3-months and a post-assessment at 6-months.
  Interventions: Other: Blood Pressure Technology System E

INTERVENTIONS:
Other: Blood Pressure Technology System M — Participants will be provided the blood pressure technology system M. The study staff will teach the participants how to use the system on their personal cell phones with instruction guides. Participants will be asked to use the system for 6-months.
  Arms: Blood Pressure Technology System M
Other: Blood Pressure Technology System E — Participants will be provided the blood pressure technology system E. The study staff will teach the participants how to use the system on their personal cell phones with instruction guides. Participants will be asked to use the system for 6-months.
  Arms: Blood Pressure Technology System E

SUMMARY:
This randomized controlled trial will assess the efficacy and scalability of a blood pressure technology system intervention. The investigators will enroll 224 older adults with hypertension to identify those who are nonadherent for one hypertension medication. The participants will be randomized to one of two groups (112 per group) to use the blood pressure system for 6-months. Both groups receive information about high blood pressure and medications. One group will also receive strategies that can be used to take medications and manage blood pressure. Both groups will complete a mid-assessment at 3-months and a post-assessment at 6-months.

ELIGIBILITY:
Inclusion Criteria:

* age 65 years or older
* self-manage at least one hypertension medication
* able to read and speak English
* willing to participate in the study for six months
* currently have and use an Apple iPhone
* have hypertension medication adherence ≤ 90% in the last 2 weeks of the 4-week baseline monitoring period using an AARDEX MEMS® cap

Exclusion Criteria:

* have inadequate visual acuity (worse than 20/50 corrected near vision on Snellen test)
* experience severe depression (> 11 on Geriatric Depression Scale Short Form, GDS-15)
* are at risk for cognitive impairment (< 23 on Montreal Cognitive Assessment, MoCA)
* been instructed by their healthcare provider to withhold their blood pressure medication

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
adherence | Baseline, 3-months, 6-months
  Change in adherence (both objective and subjective) after 6 months of M system engagement versus E system use. Objective adherence is measured by Aardex Medication Event Monitoring System (MEMS). Subjective adherence is measured by the five-item Medication Adherence Report Scale (MARS-5). MARS-5 total score ranges between 5 and 25, with higher scores indicating better adherence.

SECONDARY OUTCOMES:
systolic blood pressure (BP) | Baseline, 3-months, 6-months
  6-month change in mean seated systolic BP among M system users versus E system users.
perceived competence | Baseline, 3-months, 6-months
  6-month change in perceived competence among M system users versus E system users. The four-item Perceived Competence Scale (PCS) is used to measure self-determination competence. PCS total score ranges between 4 and 28, with higher scores indicating higher perceived competence with medication adherence.
perceived autonomy | Baseline, 3-months, 6-months
  6-month change in perceived autonomy among M system users versus E system users. The Treatment Self-Regulation Questionnaire (TSRQ) is used to measure individual differences in the types of motivation or regulation. Each of the 15 questionnaire items represents a reason for engaging in or changing a health behavior. Responses use a seven-point scale ranging from 1 (not at all true) to 7 (very true). Higher numbers indicate higher autonomous motivation, controlled motivation, or amotivation.
mobile device proficiency | Baseline, 3-months, 6-months
  6-month change in mobile device proficiency among M system users versus E system users. Proficiency is measured with the Mobile Device Proficiency Questionnaire (MDPQ-16). The MDPQ-16 total score ranges from 8 to 40, with higher scores reflecting greater proficiency.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Arizona, Tucson, Arizona
  - University of Illinois Urbana-Champaign, Champaign, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Data and resources generated during the performance of the project will be shared with the research community primarily via conference presentations, journal articles, and summary reports made available on laboratory and company websites. Technical manuals created during the project may be made publicly available via websites geared towards sharing resources in the research community or licensed, as appropriate, and after University review. Completely de-identified final data will be shared with existing and new collaborators of the laboratories participating in the project and with new collaborators who may initiate contact by emailing one of the PIs, using HIPAA-compliant file transfer methods once the investigators complete a data-sharing agreement. The data-sharing agreement will ensure that privacy, confidentiality standards, and data security will be maintained at the recipient site and will prohibit manipulation of data

REFERENCES:
- [Background] Chan AHY, Horne R, Hankins M, Chisari C. The Medication Adherence Report Scale: A measurement tool for eliciting patients' reports of nonadherence. Br J Clin Pharmacol. 2020 Jul;86(7):1281-1288. doi: 10.1111/bcp.14193. Epub 2020 May 18. PMID 31823381
- [Background] Williams GC, Freedman ZR, Deci EL. Supporting autonomy to motivate patients with diabetes for glucose control. Diabetes Care. 1998 Oct;21(10):1644-51. doi: 10.2337/diacare.21.10.1644. PMID 9773724
- [Background] Roque NA, Boot WR. A New Tool for Assessing Mobile Device Proficiency in Older Adults: The Mobile Device Proficiency Questionnaire. J Appl Gerontol. 2018 Feb;37(2):131-156. doi: 10.1177/0733464816642582. Epub 2016 Apr 11. PMID 27255686
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Hypertension. 2018 Jun;71(6):e13-e115. doi: 10.1161/HYP.0000000000000065. Epub 2017 Nov 13. No abstract available. PMID 29133356
- [Background] Lee JY, Kusek JW, Greene PG, Bernhard S, Norris K, Smith D, Wilkening B, Wright JT Jr. Assessing medication adherence by pill count and electronic monitoring in the African American Study of Kidney Disease and Hypertension (AASK) Pilot Study. Am J Hypertens. 1996 Aug;9(8):719-25. doi: 10.1016/0895-7061(96)00056-8. PMID 8862216